CLINICAL TRIAL: NCT03960437
Title: The Effect of Etelcalcetide on Bone-tissue Properties and Calcification Propensity in End Stage Kidney Disease
Brief Title: The Effect of Etelcalcetide on CKD-MBD
Acronym: Parsabiv-MBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Nickolas, MD MS (Other)
Responsible Party: Sponsor-Investigator, Thomas Nickolas, MD MS, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6244
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease Mineral and Bone Disorder; Renal Osteodystrophy; Vascular Calcification; Hyperparathyroidism; Secondary, Renal
Keywords: Kidney disease; Bone disease; Etelcalcetide; Parsabiv
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Vascular Calcification; Hyperparathyroidism; Neoplasm Metastasis; Kidney Diseases; Bone Diseases | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Participant (Other): Every study participant will receive etelcalcetide prescribed by their treating physician for the duration of the study.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously at the end of each dialysis session. Dosing ranges from 5 mg to 15 mg set by the patient's physician.
  Other Names: Parsabiv

SUMMARY:
The proposed study will investigate the effects of etelcalcetide on the bone and blood-vessel health in patients with CKD-MBD. The investigators will test if etelcalcetide makes bone and blood-vessels healthier. The study hypotheses are that are that etelcalcetide keeps bones strong and lowers the risk of calcium deposits in blood vessels. In Aim 1, the investigators will test if 9-months of treatment with etelcalcetide improves bone strength in twenty ESKD patients with hyperparathyroidism (HPT) by bone biopsy. In Aim 2, the investigators will test if 9-months of treatment with etelcalcetide decreases serum propensity to calcify blood vessels. The potential significance of this study is to provide first-time data on the ability of etelcalcetide to protect bone and blood-vessel health in patients with ESKD.

DETAILED DESCRIPTION:
Chronic kidney disease - mineral and bone disease (CKD-MBD) is a disorder of bone and mineral metabolism in patients with CKD. When kidney function is poor, levels of vitamin D, phosphate and parathyroid hormone become abnormal and patients are at risk for bone disease and fractures (renal osteodystrophy) and the deposition of calcium in blood vessels and muscles. CKD-MBD increases the risk of fractures, heart attacks, strokes, and death. Treatment of CKD-MBD is focused on lowering levels of parathyroid hormone (PTH) by giving vitamin D and lowering levels of phosphorous by giving phosphate binders. In patients with end stage kidney disease (ESKD), target levels of PTH recommended by the Kidney Disease Improving Global Outcomes (KDIGO) guidelines are in the range of 2-9 times the upper limit of normal (ULN) for the PTH assay. In many cases, in patients with long-standing ESKD, the parathyroid gland may no longer respond to treatment with vitamin D and phosphate lowering. In these cases, treatment with a calcimimetic, a medicine that increases the sensitivity of the parathyroid gland to serum levels of calcium, can restore PTH levels to goal.

ELIGIBILITY:
Inclusion Criteria:

For All Aims:

1. Patient has provided informed consent.
2. Patient is 18 years of age or older.
3. Patient must be receiving maintenance hemodialysis for at least 3 months, with adequate hemodialysis with a delivered Kt/V 1.2 or urea reduction ratio (URR) 65% within 4 weeks prior to screening laboratory assessments.
4. Dialysate calcium concentration must be stable for at least 4 weeks prior to screening laboratory assessments.
5. Patient must have severe HPT as defined by two laboratory screening pre-dialysis serum PTH values >9-times ULN for the PTH assay, measured on two consecutive monthly lab checks prior to entering the study.
6. The patient has an uncontrolled PTH defined by KDIGO as a PTH greater than 9 times the upper limit of normal of the assay (720 pg/mL for Rogosin):

   AND one of the following:
   * The patient has never been on cinacalcet OR,
   * The patient received daily cinacalcet for less than 3 months and has been off cinacalcet for at least 3 months prior to enrollment OR ,
   * The patient received daily cinacalcet for more than 3 months and has been off cinacalcet for at least 6 months prior to enrollment OR,
   * The patient received a modified dose of three times weekly cinacalcet and has been off cinacalcet for at least one month prior to enrollment.
7. Scheduled to receive etelcalcetide for the treatment of HPT per standard of care.
8. If receiving vitamin D sterols, patient must have had no more than a maximum dose change of 50% within the 4 weeks prior to screening laboratory assessments, remain stable through randomization, and be expected to maintain stable doses for the duration of the study, except for adjustments allowed per protocol*.
9. Patient must have one screening pre-dialysis serum Ca laboratory value at least at the lower limit of normal for the assay measured within 4 weeks prior to entering the study.
10. A patient receiving calcium supplements must have had no more than a maximum dose change of 50% within 2 weeks prior to screening laboratory assessments and remain stable throughout the study, except for adjustments allowed per protocol*.
11. A patient receiving phosphate binders must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening laboratory assessments, remain stable through, and be expected to maintain stable dose for the duration of the study, except for adjustments allowed per protocol*.
12. The treating physician considers the etelcalcetide dose and timing points described in this protocol as acceptable/optimal for their patient.
13. Female patients must be willing to use highly effective contraception during the study and for 3 months after the last dose of etelcalcetide (unless postmenopausal or surgically sterilized).

For Aim 1:

1. Total alkaline phosphatase ≥ the upper tertile of the reference range for the assay

Exclusion Criteria:

For All Aims:

1. Currently receiving treatment in an investigational device or drug study, or less than 30 days since ending treatment on an investigational device or drug study(s).
2. Currently receiving investigational procedures while participating in this study.
3. Patient with controlled PTH as defined by KDIGO as a PTH of 2 to 9 times the upper limit of normal of the assay.
4. Patients has received a bisphosphonate, denosumab or teriparatide during the 12 months prior to screening.
5. Anticipated or scheduled parathyroidectomy during the study period.
6. Patient has received a parathyroidectomy within 6 months prior to dosing.
7. Scheduled kidney transplant during the study period or anticipated living donor evaluation within three months of recruitment
8. Patient has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator.
9. Bilateral lower extremity amputations or non-ambulatory
10. Metabolic bone diseases not related to the kidney (i.e., Pagets, Osteogenesis Imprefecta)
11. Untreated hyperthyroidism or hypoparathyroidism
12. Malignancy within the last 5 years (except non-melanoma skin cancers or cervical carcinoma in situ).
13. Patient is pregnant or nursing.
14. Patient likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the patient and Investigator's knowledge.
15. Weight >300 pounds

For Aim 1 (Bone biopsy):

1. Allergy to tetracycline or demeclocycline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nickolas, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Khairallah P, Cherasard J, Sung J, Agarwal S, Aponte MA, Bucovsky M, Fusaro M, Silberzweig J, Frumkin GN, El Hachem K, Schulman L, McMahon D, Allen MR, Metzger CE, Surowiec RK, Wallace J, Nickolas TL. Changes in Bone Quality after Treatment with Etelcalcetide. Clin J Am Soc Nephrol. 2023 Nov 1;18(11):1456-1465. doi: 10.2215/CJN.0000000000000254. Epub 2023 Aug 14. PMID 37574661

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Participant
Started | 22
Completed | 13
Not Completed | 9
Not completed — Removed by PI | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Participant
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Washout of Cinacalcet Required [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in PTH Levels
Description: Mean percent change in parathyroid hormone (PTH) levels will be calculated.
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the study
Measure: Mean (Standard Error); unit: percentage of change in PTH levels
Arm/Group | Study Participant
Number analyzed (Participants) | 13
percentage of change in PTH levels
  Baseline | 0 (0)
  6 months | -54.14 (11.50)
  9 months | -64.04 (8.62)

2. Primary Outcome: Change in Bone Mineral Density (BMD) of the Femoral Neck by Dual-energy X-ray Absorptiometry (DXA)
Description: To test if 9-months of treatment with etelcalcetide changes femoral neck areal BMD, a change in age and sex adjusted Z-Score will be calculated from baseline to 9 months. A Z-Score of zero represent the population mean and higher Z-Scores indicate a better outcome.
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the study.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Study Participant
Number analyzed (Participants) | 13
Z-score | 0.43 (0.1)

3. Primary Outcome: Propensity as Measured by T50
Description: The propensity to calcify soft tissues will be measured by T50 for 9 months of treatment. T50 is a novel serum-based marker that assesses the propensity of calcification in serum. Shorter T50 indicates greater propensity to calcify.
Time Frame: 9 months
Population: No data, as measured by T50, was collected. Therefore there is no data that can be reported.
Arm/Group | Study Participant
Number analyzed (Participants) | 0

4. Primary Outcome: Percent Change in Mean Hardness
Description: Hardness will be measured by Ramen nano-indentation and mineralization measured by histomorphometry obtained (in GPa).
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the histomorphometry.
Measure: Mean (Standard Error); unit: percent of change in hardness
Arm/Group | Study Participant
Number analyzed (Participants) | 5
percent of change in hardness | 2.68 (8.92)

5. Secondary Outcome: Change in Bone Mineral Density (BMD) of the Spine by DXA
Description: To test if 9-months of treatment with etelcalcetide improves spine BMD, a change in age and sex adjusted Z-Score will be calculated from baseline to 9 months. A Z-Score of zero represent the population mean and higher Z-Scores indicate a better outcome.
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the study.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Study Participant
Number analyzed (Participants) | 13
Z-score | 0.27 (0.1)

6. Secondary Outcome: Change in Bone Mineral Density (BMD) of Total Hip by DXA
Description: To test if 9-months of treatment with etelcalcetide improves total hip BMD, the change in age and sex adjusted Z-Score will be calculated from baseline to 9 months. A Z-Score of zero represent the population mean and higher Z-Scores indicate a better outcome.
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the study.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Study Participant
Number analyzed (Participants) | 13
Z-score | 0.12 (0.07)

7. Secondary Outcome: Change in Bone Formation Rate
Description: A quadruple label method will be used to assess effects of etelcalcetide on the bone formation rate. A tetracycline double label will be used pre-etelcalcetide and a declomycin double label will be used post-etelcalcetide in a protocol that administers label 3-days on, 12-days interlude, 3-days on. A single bone biopsy will be performed 1 to 10 days after completion of the second double label. Biopsy cores will be placed into 70% ethanol then serially dehydrated and embedded in methyl methacrylate. Four-micron thick sections will be cut and left unstained for dynamic histomorphometry. A region of interest including all trabecular bone and excluding cortical bone will be analyzed separately for each tetracycline or declomycin label. Standard analysis techniques will be used to measure single, double and no labelled surfaces and distances between the two labels of each fluorescence. Standard calculations of the bone formation rate/bone surface (um3/um2/year) will be made.
Time Frame: Baseline and 9 months
Population: Only includes participants who completed the bone biopsy substudy.
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Study Participant
Number analyzed (Participants) | 5
percentage of change | -84 (17)

ADVERSE EVENTS:
Time Frame: 9 months after baseline
Arm/Group | Study Participant
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participant (N=22)
COVID-19 infection (Infections and infestations) | 1 (1)
Cardiac Event (Cardiac disorders) | 1 (1) — Cardiac event was experienced during an AVF revision under anesthesia.
Vertigo/Dizziness (General disorders) | 1 (1) — Subject was hospitalized for 2 weeks for vertigo/dizziness.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participant (N=22)
Cold Sores (Infections and infestations) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03960437/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03960437/ICF_001.pdf